CLINICAL TRIAL: NCT05691218
Title: Early High-flow Oxygen Therapy With nebuLized Beta-2-agonist Using a Vibrating Mesh for the Management of Moderate to Severe Asthma Exacerbation in the Emergency Department
Acronym: EOLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EOLE
Record Dates: First submitted 2023-01-11; First posted 2023-01-19 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Moderate Asthma Exacerbation; Severe Asthma Exacerbation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control - Standard Nebulization (Active Comparator)
  Interventions: Device: Standard Nebulization
- A-Vibrating mesh Nebulization (Experimental)
  Interventions: Device: A - Vibrating mesh nebulization
- B-Vibrating mesh Nebulization and High-flow nasal cannula heated and humidified oxygen (Experimental)
  Interventions: Device: B - Vibrating mesh nebulisation and high-flow nasal cannula heated and humidified oxygen

INTERVENTIONS:
Device: Standard Nebulization — Beta-2 adrenergic agonist administred by standrad nebulization
  Arms: Control - Standard Nebulization
Device: A - Vibrating mesh nebulization — Beta-2 adrenergic agonist nebulisation using a vibrating mesh nebuliser device (Aerogen, Galway, Ireland). Nebulisation will take place under medical air at 6L/min or medical O2 at 6L/min depending on the patient's needs and for a SpO2 target between 94-96%
  Arms: A-Vibrating mesh Nebulization
Device: B - Vibrating mesh nebulisation and high-flow nasal cannula heated and humidified oxygen — High-flow nasal cannula heated and humidified oxygen (HFNO) and nebulisation of beta-adrenergic agonist using a vibrating mesh device.
  HFNO will be administered using an Airvo2 device and beta-2 adrenergic agonist nebulisation enabled by the use of a dedicated heated humidifier and an adaptable vibrating mesh nebuliser device
  Arms: B-Vibrating mesh Nebulization and High-flow nasal cannula heated and humidified oxygen

SUMMARY:
Acute exacerbation of asthma represents an acute or sub-acute worsening in symptoms and lung function in patients with asthma. It is characterized by a progressive increase in symptoms of shortness of breath, cough, wheezing, or chest tightness. It is a common diagnosis in patients admitted in an Emergency Department for dyspnoea. Near 10 to 15% of respiratory symptoms in an ED are related to acute exacerbation of asthma.

Treatment of acute exacerbation of asthma associates nebulized beta-2 agonist adrenergic with or without ipratropium bromide, oral corticosteroids and controlled oxygen therapy to maintain SpO2 between 93 and 95%. Treatment in the ED did not vary during last years, including for patients with a lack of efficacy after first line treatment, and exacerbation are always associated with a hospitalisation in 40% of adult patients and with mortality in 1% of hospitalized patients.

Vibrating mesh nebulizers are devices using vibration to push drug through the mesh, resulting in the drug nebulization. Vibrating mesh nebulizers have been associated with better pulmonary drug delivery than jet-nebulizers, provide faster improvement in peak expiratory flow and have been associated in retrospective studies with patient prognosis, particularly in terms of throughput time and need for hospitalisation. However, no studies have prospectively compared nebulisation with a vibrating membrane device with standard nebulisation in patients with asthma exacerbation on clinically relevant criteria. Nebulisation with a vibrating membrane device may potentiate the clinical efficacy of short-acting bronchodilators, result in faster and more effective clinical improvement, and be associated with improved short- and medium-term patient outcomes.

High-flow nasal cannula heated, and humidified oxygen (HNFO) is a ventilatory support which is commonly used for the management of acute respiratory failure for acute respiratory failure in intensive care units and in emergency departments. HFNO delivers high fraction of inspired oxygen (FiO2), generates a low level of positive pressure and provides washout of dead space in the upper airways, thereby improving mechanical pulmonary properties and unloading inspiratory muscles during ARF. Consequently, HFNO is associated with a decrease in the work of breathing. During asthma exacerbation, HFNO was associated with an improvement in the dyspnea level and in the respiratory rate compared with conventional oxygen therapy. However, HFNO has never been assessed in association with nebulized beta-2 adrenergic agonist.

To resume, beta-2 adrenergic agonist nebulization with a vibrating mesh nebulizer seems effective, especially compared to standard jet nebulization. In addition, HFNO is a technique that appears to be suitable for the pathophysiological conditions of chronic reversible respiratory failure, and can be used during exacerbations of asthmatic disease. The high flow rate of gas makes it possible to control the FiO2 in order to avoid hyperoxia, to generate a PEEP effect, to reduce the patient's work of breathing and the respiratory resistance, and to avoid the re-inhalation of CO2 by a dead space wash-out.

In the EOLE study, the investigators propose to compare three therapeutic management strategies. One standard strategy (nebulisation with a jet-nebulizer), and two experimental strategies (nebulisation with a vibrating mesh device, and nebulisation with a vibrating mesh device in association with HFNO).

The investigators hypothesise that bronchodilator nebulization with a vibrating mesh nebulizer is more effective than jet-nebulizers for the management of patients admitted for asthma exacerbation and non-responders or with lack to efficacy to initial treatment. Furthermore, the investigators also hypothesise that the addition of the physiological effects of HFNO may enhance the efficacy of the treatment.

The therapeutic effects of nebulisation with a vibrating membrane device alone or with the addition of the physiological effects of HFNO could constitute a new approach to the management of asthma patients, particularly in patients who are insufficiently responsive or non-respondent to initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or over 18 years
* admitted in an Emergency Department with a clinical suspicion of acute exacerbation of asthma according to the Global Initiative for Asthma (GINA) criteria.
* with at least one of the following criteria 60mn after a first treatment by beta-2 agonist adrenergic nebulization with 3 x 5 mg of terbutaline:

  * Respiratory rate over 22 breaths/min
  * Peak flow < 50% of predictive normal value
  * SpO2 < 95% in room air
  * Signs of severe asthma exacerbation (at least one criteria):

Talks in word, Agitation, Sits hunched forwards, Accessory muscles in use

* Free subject, without guardianship or curatorship or subordination
* Patients benefiting from a Social Security scheme or benefiting from it through a third party
* Informed consent signed by the patient after clear and honest information about the study

Exclusion Criteria:

* Acute exacerbation of asthma during the last 30 days
* Clinical suspicion of acute exacerbation of asthma due to anaphylaxis, pneumothorax, pneumomediastinum, pneumonia or atelectasis.
* At least ONE of the following serious signs: drowsiness, confusion, auscultatory silence
* Clinical suspicion of another pathology that could explain the respiratory failure such as heart failure, laryngeal obstruction, pulmonary embolism, etc
* Patients with neurological (Glasgow < 13) or hemodynamical failure (Mean Arterial Pressure < 65 mmHg)
* contraindication to treatment with a beta-2-adrenergic agonist
* History of hypersensitivity (allergy) to terbutaline or any of the constituents
* Contraindication to OHD
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, people assessed GIR1 or GIR 2 (AGGIR grid), adults under legal protection
* Pregnant or breastfeeding women, Women at age to procreate and not using effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Number of responding patients one hour after inclusion | 1 hour
  A responding patient is defined by a patient responding to all the following criteria :
  * Respiratory rate ≤ 22 ventilations /minutes
  * Peak flow > 60% of theorics
  * SpO2 ≥ 95% in room air
  * Absence of clinical signs related with severe exacerbation of asthma

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MARJANOVIC, MD PHD, Principal Investigator — CHU Poitiers
Locations (1):
- University Hospital of Poitiers, Poitiers, France, France